CLINICAL TRIAL: NCT04188795
Title: Evaluation of the Effectiveness of Delirium Preventive Care Protocol for Hip Fracture Patients
Brief Title: Evaluation of the Effectiveness of Delirium Preventive Care Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 50687469-2244
Record Dates: First submitted 2019-11-20; First posted 2019-12-06 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2019-11

CONDITIONS: Delirium
Keywords: Care protocol; Delirium; Nursing care; Hip fracture
MeSH Terms: conditions — Delirium; Hip Fractures

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial conducted at Gulhane Training and Research Hospital , Orthopedic and Traumatologic clinic between May 2018 and January 2019.The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomized controlled trials (RCTs) has been used to describe the methods.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who met the criteria for inclusion in the study and volunteered to participate in the study were divided into experimental and control groups by block randomization method.
  After obtaining written informed consent, the Patient Information Form, Mini Nutritional Assessment- Short Form, Confusion Assessment Method, Barthel Index and Visual Analog Scale were applied to patients. Nursing care was applied to hip fracture patients in the experimental group in accordance with the care protocol developed to prevent delirium. Delirium preventive care protocol was consist of; psychosocial care, monitoring of oxygen saturation, prevention of dehydration, nutritional support, normal elimination, pain control, sleep regulation, avoidance of bladder catheterization and early mobilization.
  Confusion Assessment Method, Barthel Index and Richards-Campbell Sleep Questionnaire were repeated to patients on the first postoperative day and on the third day.
  Interventions: Procedure: Delirium Preventive Care Protocol
- Control Group (No Intervention): After obtaining written informed consent, the Patient Information Form, Mini Nutritional Assessment- Short Form, Confusion Assessment Method, Barthel Index and Visual Analog Scale were applied to patients. Routine nursing care was applied to hip fracture patients in the control group. Confusion Assessment Method, Barthel Index and Richards-Campbell Sleep Questionnaire were repeated to patients on the first postoperative day and on the third day.

INTERVENTIONS:
Procedure: Delirium Preventive Care Protocol — Nursing care was applied to hip fracture patients in the experimental group in accordance with the care protocol developed to prevent delirium. Delirium preventive care protocol was consist of; psychosocial care, monitoring of oxygen saturation, prevention of dehydration, nutritional support, normal elimination, pain control, sleep regulation, avoidance of bladder catheterization and early mobilization.
  Confusion Assessment Method, Barthel Index and Richards-Campbell Sleep Questionnaire were repeated to patients on the first postoperative day and on the third day.
  Arms: Intervention

SUMMARY:
The prospective, randomized controlled experimental trial investigates the effectiveness of delirium preventive care protocol for hip fracture patients.

DETAILED DESCRIPTION:
The aim of this prospective, randomized controlled experimental trial is to evaluate the effectiveness of delirium preventive care protocol on pain, functional status, sleep quality and delirium prevention in patients with hip fracture.

This research was conducted at a training and research hospital's orthopedics and traumatology department. The study sample was compromised of 80 patients with hip fracture. Intervention and control groups were applied after block randomization. Study data was collected by using Patient Information Form, Mini-Cog Test, Confusion Assessment Method, Visual Analogue Scale, Barthel Index, Mini Nutritional Assessment-Short Form and Richards Campbell Sleep Questionnaire. The patients in the intervention group were provided with nursing care in accordance with the delirium preventive care protocol developed with the support of literature. In the control group, routine nursing care was provided in line with the clinical procedure. The data was analyzed by using number, percentage, mean, standard deviation, median, Interquartile Range, Student's t test, Mann-Whitney U test, Pearson's chi square test, Fisher corrected chi-square test, ANOVA test, Paired Sample t test, Friedman test, Wilcoxon test and Cronbach α coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery for hip fracture,
* 65 years and older,
* No communication problems in Turkish,
* Without cognitive impairment,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Patients who could not be evaluated by the investigator before the operation
* Patients with dementia and Mini-Cog test less than 3 points
* Patients with a history of cerebrovascular accident
* Patients with severe comorbidity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire (RCSQ) | 4 minutes.
  It was applied to patients at first admission to the clinic, on the first and third postoperative day. The scale developed by Richards in 1987; It consists of six items that assess the depth of night's sleep, the time to fall asleep, the frequency of waking up, the time to wake up, the quality of sleep and the noise level in the environment. Each item is evaluated on the chart from 0 to 100. A score of 0-25 indicates a very poor sleep and a score of '76 -100 indicates a very good sleep. The higher the scale score, the better the sleep quality of the patients.
  The total sleep score is calculated by taking the average of the depth of sleep, the time to fall asleep, the frequency of waking up, the time to stay awake and the quality of sleep.
Barthel Index (BI) | 5 minutes.
  Patients filled at frst admission to the clinic, on the first and third postoperative day was developed in 1965 by Mahoney and Barthel. It is used to determine the level of independence of individuals in their activities. The Barthel Index measures the social and physical function of daily life and consists of 10 items that assess the individual's ability to meet daily functions (nutrition, bathing, personal care, dressing, toileting, mobility on flat surfaces, transfer, climbing stairs, bowel and bladder function) without assistance. Each item is scored between 0-15 (varies according to the question). Barthel Index total scores vary between 0-100; 0-20 points completely addiction; 21-61 points severe addiction; Moderate dependence of 62-90 points; 91-99 points mild addiction; 100 points explain independence. In the studies using the Barthel Index, 60 points were taken as the limit and scores above 60 explain the ability to function independently.
Visual Analog Scale (VAS) | 1 minute.
  It was applied to patients at first admission to the clinic, on the first and third postoperative day. It is used to measure the severity of pain. It is easy to use and the same in every language. At the two ends of a ten-centimeter line, two end definitions of the parameter to be evaluated are written and the patient is asked to indicate where his or her condition is appropriate by drawing a line or by pointing or pointing (0: I have no pain, 10: I have unbearable pain). The length of the distance from the absence of pain to the location of the patient indicates the pain of the patient. Less than three of this numerical expression indicates mild pain, three to seven indicates moderate pain, and more than seven indicates severe pain.
Mini Nutritional Assesment- Short Form (MNA-SF) | 2 minutes.
  It was applied to patients at first admission to the clinic for evaluating of malnutrition. Its use in the elderly is recommended by the European Society for Clinical Nutrition and Metabolism (ESPEN). According to the screening score; 0-7 points indicate malnutrition, 8-11 points indicate malnutrition risk, 12-14 points indicate normal nutritional status.

OTHER OUTCOMES:
Confusion Assessment Method- Intensive Care Unit (CAM-ICU) | 5 minutes.
  It was applied to patients at first admission to the clinic, on the first and third postoperative day and in cases of change of consciousness. The scale was developed by Ely et al in 2001. The scale consists of four items. In the first item, sudden changes in consciousness or fluctuation; In the second article, squeezing the hand with letter A in less than 12 in the attention assessment test tests the two most important signs of delirium, fluctuations in the level of consciousness and distortion of attention. In the third article, it is evaluated whether the thought organization is disrupted or not by four questions and a simple command. The fourth item is related to the assessment of consciousness level. According to this scale, the first two items and one of the third or fourth items must be positive for the diagnosis of delirium. CAM-ICU, which is the most widely used scale that best complies with Diagnostic and Statistical Manual of Mental Disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten Guvenc, Proffessor, Study Director — University of Health Sciences, Gulhane Faculty of Nursing
Locations (3):
- Turkey (Türkiye) (3):
  - University of Heath Sciences, Gulhane Faculty of Nursing, Ankara
  - University of Health Sciences, Faculty of Nursing, Ankara
  - University of Health Sciences, Gulhane Faculty of Nursing, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durst J, Wilson D. Effects of protocol on prevention of delirium in hospitalized hip fracture patients: A quality improvement project. Int J Orthop Trauma Nurs. 2020 Feb;36:100710. doi: 10.1016/j.ijotn.2019.100710. Epub 2019 Aug 1. PMID 31521618
- [Background] Holly C. Primary Prevention to Maintain Cognition and Prevent Acute Delirium Following Orthopaedic Surgery. Orthop Nurs. 2019 Jul/Aug;38(4):244-250. doi: 10.1097/NOR.0000000000000569. PMID 31343628
- [Background] Prestmo A, Hagen G, Sletvold O, Helbostad JL, Thingstad P, Taraldsen K, Lydersen S, Halsteinli V, Saltnes T, Lamb SE, Johnsen LG, Saltvedt I. Comprehensive geriatric care for patients with hip fractures: a prospective, randomised, controlled trial. Lancet. 2015 Apr 25;385(9978):1623-33. doi: 10.1016/S0140-6736(14)62409-0. Epub 2015 Feb 5. PMID 25662415
- [Background] Flikweert ER, Izaks GJ, Knobben BA, Stevens M, Wendt K. The development of a comprehensive multidisciplinary care pathway for patients with a hip fracture: design and results of a clinical trial. BMC Musculoskelet Disord. 2014 May 30;15:188. doi: 10.1186/1471-2474-15-188. PMID 24885674
- [Background] Marcantonio ER, Flacker JM, Wright RJ, Resnick NM. Reducing delirium after hip fracture: a randomized trial. J Am Geriatr Soc. 2001 May;49(5):516-22. doi: 10.1046/j.1532-5415.2001.49108.x. PMID 11380742
- [Derived] Unal N, Guvenc G, Naharci M. Evaluation of the effectiveness of delirium prevention care protocol for the patients with hip fracture: A randomised controlled study. J Clin Nurs. 2022 Apr;31(7-8):1082-1094. doi: 10.1111/jocn.15973. Epub 2021 Jul 23. PMID 34302312

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT04188795/Prot_SAP_000.pdf